CLINICAL TRIAL: NCT06239818
Title: Assessing the Effects of Photobiomodulation on Clinical Recovery From Concussion in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: TIRR/Mission Connect (Other)
Responsible Party: Principal Investigator, Summer Ott, Psy.D., Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-23-0871
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Sports-related Concussion
MeSH Terms: interventions — Low-Level Light Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment: Photobiomodulation therapy (PBMt) (Experimental)
  Interventions: Device: Photobiomodulation therapy (PBMt); Other: Standard of Care
- Control (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Photobiomodulation therapy (PBMt) — Participants will be asked to use the photobiomodulation (PBM) device for 20 minutes, daily (e.g., Monday - Sunday) for a total of 30 days. The device will be preprogrammed and automatically switched off after 20 minutes.
  Arms: Treatment: Photobiomodulation therapy (PBMt)
Other: Standard of Care — The patient is provided with verbal and written education including what a mild traumatic brain injury (mTBI) is, favorable expectations for recovery, and advice about how to manage specific symptoms. Relative rest for the first 24-48 hours after an mTBI is recommended as the main goal is to alleviate symptoms and reduce demands on the brain. After an initial period of relative rest and symptom stabilization, patients are encouraged to gradually resume normal daily activities as tolerated. Physical and cognitive activities can be progressively resumed at a pace that does not worse existing or create new symptoms. Education, return to activity advice, and symptom management are all reviewed in subsequent visits as needed.

SUMMARY:
The purpose of this study is to compare effects of Photobiomodulation therapy (PBMt) to standard of care in adolescent athletes at risk for delayed recovery from subacute sports concussion, to substantiate the impact of subacute PBMt over time on functional and structural connectivity of the brain using advanced MRI sequences and to correlate the psychological and behavioral outcomes to neuroimaging findings

ELIGIBILITY:
Inclusion Criteria:

* current participants in a school- or club-sponsored sport (contact or non-contact)
* access to wireless internet service at home
* diagnosis of sports-related concussion (SRC) (according to consensus diagnostic criteria) by a licensed healthcare provider,3-7 days from the concussive injury at the time of enrolment
* considered at-risk for protracted recovery based on Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) performance and symptom reporting on the Post-Concussion Symptom Scale (PCSS)

Exclusion Criteria:

* acute neurologic deterioration to a Glasgow Coma Scale score less than 13
* neurosurgical intervention
* abnormal CT scan
* concomitant extracranial injury worse than mild
* pre-injury conditions which confound effects of SRC (e.g., epilepsy, schizophrenia, bipolar illness, mental deficiency, hospitalization for TBI)
* substance dependence
* inability to speak fluent English
* Individuals who are taking benzodiazepines, anti-convulsants, mood stabilizers, stimulants, opioids, sleep aids, or other neuropsychiatric medications

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in depression as assessed by the Neuro-QoL Short Form v1.1 - Pediatric Depression scale | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  This is an 8 item questionnaire, and each item is scored on a 5 point Likert scale from 1 (never) to 5 (almost always), for a total score range of 8 to 40 and with a higher score indicating a worse outcome.
Change in anxiety as assessed by the Neuro-QoL Short Form v1.0 - Pediatric Anxiety scale | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  This is an 8 item questionnaire, and each item is scored on a 5 point Likert scale from 1 (never) to 5 (almost always), for a total score range of 8 to 40 and with a higher score indicating a worse outcome.
Change in intensity of post-concussion symptoms as assessed by Total Symptom Score on the Post-Concussion Symptoms Scale (PCSS) of the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  The PCSS of the ImPACT Concussion Test consists of a list of 22 symptoms for which participants rate the intensity of a symptom from 0 (none) to 6 (severe), for a Total Symptom Score range of 0 to 132 and with a higher score indicating a higher symptom total.
Change in quality of sleep as assessed by the Adolescent Sleep-Wake Scale-S (ASWS-Short Version) | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  The Total Sleep Quality Score will be reported, and it ranges from 1 to 6. A higher score indicates better sleep quality.
Change in brain volume as assessed by Magnetic Resonance Imaging (MRI) of the brain | Baseline (3-7 days post injury), Visit 3 (30 days post injury)
Change in Diffusion Tensor Image Analysis Along the Perivascular Space (DTI-ALPS) as assessed by MRI of the brain | Baseline (3-7 days post injury), Visit 3 (30 days post injury)
Change in Fractional Anisotropy (FA) of compact white matter as assessed by MRI of the brain | Baseline (3-7 days post injury), Visit 3 (30 days post injury)
Change in Radial Diffusivity (RD) of compact white matter as assessed by MRI of the brain | Baseline (3-7 days post injury), Visit 3 (30 days post injury)

SECONDARY OUTCOMES:
Change in cognitive function as assessed by composite score on the Verbal Memory component of the ImPACT Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  Composite score on the Verbal Memory component of the ImPACT Concussion Test will be reported, and it ranges from 0 to 100, with a higher score indicating a better outcome.
Change in cognitive function as assessed by composite score on the Visual Memory component of the ImPACT Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  Composite score on the Visual Memory component of the ImPACT Concussion Test will be reported, and it ranges from 0 to 100, with a higher score indicating a better outcome.
Change in cognitive function as assessed by composite score on the Visual Motor Speed component of the ImPACT Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  Composite score on the Visual Motor Speed component of the ImPACT Concussion Test will be reported, and it ranges from 0 to 50, with a higher score indicating a better outcome.
Change in cognitive function as assessed by composite score on the Reaction Time component of the ImPACT Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  Composite score on the Reaction Time component of the ImPACT Concussion Test will be reported, and it ranges from 0 to 1.50, with a lower time indicating a better outcome.
Change in cognitive function as assessed by composite score on the Impulse Control component of the ImPACT Concussion Test | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  Composite score on the Impulse Control component of the ImPACT Concussion Test will be reported, and it ranges from 0 to 30, with a lower score indicating a better outcome.
Change in cognitive function as assessed by the Neuro-QoL Short Form v2.0 - Pediatric Cognitive Function scale | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  This is an 8 item questionnaire, and each item is scored from 1 (very much) to 5 (not at all), for a total score range of 8 to 40 and with a higher score indicating a better outcome.
Change in stress as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Short Form v1.0 - Psychological Stress Experiences 8a scale | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  This is an 8 item questionnaire, and each item is scored from 1 (never) to 5 (always), for a total score range of 8 to 40 and with a higher score indicating more stress.
Change in quality of life as assessed by the PROMIS Pediatric Scale v1.0 - Global Health 7 scale | Baseline (3-7 days post injury), Visit 2 (10-14 days post injury), Visit 3 (30 days post injury)
  This is a 7 item questionnaire, and each item is score from 1 to 5, for a total score range of 7 to 35 and with a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Ott, PsyD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No